CLINICAL TRIAL: NCT00573963
Title: Determination of the Efficay of the Transversus Abdominis Plane (TAP) Block as Part of a Multimodal Regimen for Post-cesarean Delivery Analgesia: a Double Blinded Placebo-controlled Study.
Brief Title: Efficacy of the Transversus Abdominus Plane (TAP) Block for Post-Cesarean Delivery Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Dr. Jose C.A. Carvalho, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-11; 07-0245-A
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Pain
Keywords: Cesarean section
MeSH Terms: conditions — Pain | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Ropivacaine
  Interventions: Drug: ropivacaine
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: saline solution

INTERVENTIONS:
Drug: ropivacaine — 2 injections of 20mL 0.375% ropivacaine - one given on each side.
  Other Names: Naropin
  Arms: 1
Drug: saline solution — 2 injections of 20mL plain saline solution - one on each side.
  Arms: 2

SUMMARY:
The purpose of this study is to determine if patients having the transversus abdominal place (TAP) block at the end of a cesarean delivery have less pain in the post-delivery period than those who do not. Freezing medication is injected between the layers of muscle on either side of the belly, to freeze the nerves that carry pain stimuli from an abdominal wound. This technique has been useful for many abdominal operations, and has recently been studied in cesarean sections, however more information is needed.

DETAILED DESCRIPTION:
A cesarean section is a surgical procedure and, like all surgeries, there is pain after the operation. The purpose of this study is to find out if patients have less pain after a cesarean delivery when they receive an injection of local anesthetic on either side of their abdomen, into the plane of the transversus abdominis muscle. We are also interested in whether or not this injection decreases the need for other pain-killing medication during this time.

Patients will randomly be assigned to receive either local anesthetic or a placebo. In addition, all patients will receive the usual standard of care and medication for pain. At 6, 12, 24 and 48 hours after the operation, patients will be asked about their pain and satisfaction with pain management. The risk of side effects is very low, as the block is done in an area with low blood supply. We propose that the addition of the TAP block to the current multi-modal regimen of post-cesarean pain management will reduce pain scores and requests for additional analgesia post-operatively, as well as increase patient satisfaction with their pain control.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing elective cesarean delivery

Exclusion Criteria:

* Patients unable to communicate in English
* Patients with an American Society of Anesthesiologists (ASA) classification of 3 or higher
* Patients with contraindications to spinal anesthesia
* Patients with an allergy to ropivacaine, morphine, ketorolac or acetaminophen
* Patients who have taken any pain medication in the past 24 hours
* Patients with a BMI > 40

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Pain score by visual analogue scale (VAS) on movement at 24 hours postoperatively. | 24 hours

SECONDARY OUTCOMES:
Pain at rest and on movement by VAS at 6, 12, 24 & 48 hours postoperatively. | 48 hours
Opioid consumption at 6, 12, 24 & 48 hours postoperatively. | 48 hours
Time to first maternal request for supplemental analgesia. | 48 hours
Maternal satisfaction with pain management on a scale of 0-10, at 6, 12, 24 and 48 hours postoperatively. | 48 hours
Presence of pain 6 weeks postoperatively. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada